CLINICAL TRIAL: NCT03137641
Title: Assessment of Nurses Internal Contamination by Antineoplastic Drugs in Hospital Centers.
Brief Title: Nurses Internal Contamination by Antineoplastic Drugs.
Acronym: CACIES
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Bordeaux PharmacoEpi (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2013/30
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Antineoplastic Drugs Contamination Prevalence
Keywords: occupational exposure; antineoplastic drugs; biomonitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses in contact with chemotherapies: It is a nurses cohort, who administer chemotherapies or are in charge of patients treated by chemotherapie. Three urine samples are collected:
  first : between 0 to 3h before the beginning of the workday second : between 0 to 2h after the end of the workday third : between 7 to 10h after the end of the workday
  Interventions: Other: Nurses urine samples

INTERVENTIONS:
Other: Nurses urine samples — Collected urine samples from nurses in contact with antineoplastic drugs.

SUMMARY:
CACIES is a descriptive study conducted in two hospital centers in France to assess nurses internal contamination by antineoplastic drugs.

DETAILED DESCRIPTION:
The increase of cancer incidence contributes to a growing number of administered chemotherapies in care services. These antineoplastic drugs are not selective in their mechanisms of action, affecting noncancerous as well as cancerous cells, leading to several known side effects in treated patients. Health care professionals are increasingly exposed to antineoplastic drugs and can be potentially contaminated by these molecules. This is a key concern as part of assessment and occupational risk management in healthcare settings.

Occupational Health and Safety Department, in collaboration with Clinical and Toxicology Laboratory of university Hospital Bordeaux, developed analytical tools to assess this contamination in health care professional's urines, and the new acquisition of a high-sensitivity measurement equipment (LC-MS/MS) improved assays methods in terms of sensitivity and detection limits.

The main objective of the study is to assess internal contamination prevalence by the studied antineoplastic drugs (5-fluorouracil, cyclophosphamide, doxorubicin, ifosfamide, methotrexate) in nursing staff who administers these chemotherapies or is in charge of patients treated by these chemotherapies, in two French hospital centers: University Hospital Bordeaux and IUCT-Oncopole of Toulouse (Institut Universitaire du Cancer de Toulouse), including about fifteen services selected on their use of these specific chemotherapies.

The secondary objectives of the study are on the one hand, to describe for each of the five studied antineoplastic drugs the internal contamination prevalence in nursing staff, and concentration level associated to this contamination in contaminated nursing staff, and on the other hand, to identify contamination-associated factors in exposure characteristics and personal protective equipment use.

This is a descriptive, multicentre, transverse and prospective study.

ELIGIBILITY:
Inclusion Criteria:

* To be a nurse with Registered Nurse Licensure (IDE: Infirmier Diplômé d'Etat), practising in one of the selected services in Bordeaux teaching hospital or in IUCT-Oncopole,
* To have used at least one of the five antineoplastic drugs and/or to have cared one patient treated by one of the five antineoplastic drugs (5-fluorouracil, cyclophosphamide, doxorubicin, ifosfamide, methotrexate) in the workday of participation to the study (day with urine samples),
* To have accepted to participate to the study and signed the participation consent form.

Exclusion Criteria:

* To be a nursing student,
* To be treated or to have been treated in the year before the workday of study participation by one of the five antineoplastic drugs (5-fluorouracil, cyclophosphamide, doxorubicin, ifosfamide, methotrexate)
* To have at home, someone treated by one of the five antineoplastic drugs in the month before the workday of study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nurses working in anticancer unit.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Internal contamination by at least one antineoplastic drug. | inclusion day
  Presence or absence of internal contamination by at least one antineoplastic drug of the five studied antineoplastic drugs (5-fluorouracil, cyclophosphamide, doxorubicin, ifosfamide, methotrexate) in at least one of the three urine samples collected by subject.

SECONDARY OUTCOMES:
Nurses contamination prevalence. | inclusion day
  5 studied antineoplastic drugs concentration in urine samples.
Socio-demographic factors. | inclusion day
  Assessed by age, sexe, pregnancy, cigarette addiction questionnaire
Practical work conditions. | inclusion day
  Assessed by practical work conditions questionnaires.
Patients management treated by 5 studied antineoplastic drugs. | inclusion day
  Assessed by practical work conditions questionnaires.
Safety equipment use. | inclusion day
  Assessed by safety equipment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: PARIENTE Antoine, Pr, Study Chair — Bordeaux PharmacoEpi (BPE)
Locations (3):
- France (3):
  - Hôpital Pellegrin, Bordeaux
  - CHU de Toulouse, Toulouse
  - IUCT-Oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villa A, Molimard M, Bignon E, Martinez B, Rouyer M, Mathoulin-Pelissier S, Baldi I, Verdun-Esquer C, Canal-Raffin M. Study protocol for the assessment of nurses internal contamination by antineoplastic drugs in hospital centres: a cross-sectional multicentre descriptive study. BMJ Open. 2019 Nov 10;9(11):e033040. doi: 10.1136/bmjopen-2019-033040. PMID 31712349